CLINICAL TRIAL: NCT01296659
Title: Phase Ib Study of Oral Ridaforolimus in Combination With Standard Chemotherapy for Patients With Advanced Unresectable Soft Tissue Sarcoma
Brief Title: Study of Oral Ridaforolimus in Combination With Standard Chemotherapy for Soft Tissue Sarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator left institution.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDD 10-09
Record Dates: First submitted 2011-02-03; First posted 2011-02-15 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: sarcoma; Ridaforolimus; soft tissue sarcoma; unresectable sarcoma
MeSH Terms: conditions — Sarcoma | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIM Arm (Experimental): Ridaforolimus combined with doxorubicin/ifosfamide/mesma (AIM)
  Interventions: Drug: ridaforolimus
- TG Arm (Experimental): Ridaforolimus combined with docetaxel and gemcitabine (TG)
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — Ridaforolimus administered orally 5 days per week in combination with standard chemotherapy
  Other Names: deforolimus

SUMMARY:
Ridaforolimus has been tested in almost 2 dozen studies; however, it has not previously been tested in combination with the standard of care chemotherapy for sarcoma as this study will. We will be looking to see if Ridaforolimus given with SOC chemo (AIM or TG) is well tolerated and to determine a Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic soft tissue sarcoma with histological or cytological proven disease. No more than 2 lines of chemotherapy in the metastatic setting in the dose escalation phase, and no more than one line of prior therapy in the expansion phase.
* ECOG performance status of ≤ 1
* A minimum life expectancy > 3 months
* At least 4 weeks must have elapsed between prior investigational therapy, chemotherapy or radiotherapy and the first dose of ridaforolimus
* Adequate hematological, hepatic and renal function (hemoglobin ≥ 9g/dl, absolute neutrophil count [ANC] ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; bilirubin ≤ ULN; alkaline phosphatase ≤ 2.5 x ULN; AST, ALT ≤ 2.5 x ULN; albumin ≥ 2.5mg/dL; creatinine ≤ 1.5 x ULN)
* Serum cholesterol ≤ 350 mg/dL and triglycerides ≤400 mg/dL
* Signed informed consent
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to start of therapy and must use an approved contraceptive method as appropriate from the time of screening until 30 days after the last dose of study drug.

Exclusion Criteria:

* Uncontrolled brain metastases, spinal cord compression, or carcinomatous meningitis.
* Clinically significant unexplained bleeding within 28 days prior to entering the trial
* Uncontrolled systemic vascular hypertension
* Clinically significant cardiovascular disease
* Newly diagnosed (within 3 months of enrollment) or poorly controlled type 1 or 2 diabetes
* Have received >350 mg/m2 total dose of Doxorubicin
* Active infection requiring prescribed intervention
* Other concurrent illness
* Major surgery within 28 days before trial entry, or incompletely healed surgical incision; minor surgery or procedures within 7 days
* Previous anthracycline lifetime exposure more than 350 mg/m2 would exclude patient form AIM Arm enrollment
* Pregnant or breastfeeding
* Known allergy to macrolide antibiotics
* Concurrent treatment with medications that induce or inhibit cytochrome P450 (CYP3A).
* Known history of HIV sero-positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Define maximum tolerated dose (MTD) | 12-18 months
  Defining the maximum tolerated dose (MTD) and recommended Phase II dose for the combination ridaforolimus and SOC chemotherapy

SECONDARY OUTCOMES:
Number of Grade 2 or higher side effects with the combined therapy. | 12-18 months
  Any evidence of antitumor activity--as measured by response rate (RECIST).
Pharmacokinetics | 12-18 months
  Ridaforolimus pharmacokinetics when given in combination with SOC chemotherapy. Limited PK for SOC chemotherapy when combined with ridaforlimus. We will measure change in concentration of Ridaforolimus when combined with chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mita, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States

REFERENCES:
- See also: Cancer Therapy & Research Center's Website — http://www.ctrc.net